CLINICAL TRIAL: NCT02560207
Title: Does Continuous Cefotaxime Administration Improve Time to Attainment and Maintenance of Target Drug Levels in Critically Ill Patients?
Brief Title: Randomized Trial of Continuous Versus Intermittent Cefotaxime Infusion on ICU.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. J.G. Zijlstra, prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/468
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness | interventions — Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent cefotaxime (Active Comparator): Cefotaxime 1 gram (1000 mg) is to be administered 4 times daily for 4 days
  Interventions: Drug: Cefotaxime
- Continuous cefotaxime (Experimental): After a 1 gram (1000 mg) Cefotaxime loading dose, Cefotaxime 4 gram (4000 mg) is to be administered as a continuous infusion in 24h for 4 days .
  Interventions: Drug: Cefotaxime

INTERVENTIONS:
Drug: Cefotaxime — To assess the influence of administration route on target attainment cefotaxime is administered via two IV routes.
  Other Names: Claforan

SUMMARY:
This study evaluates target attainment after either intermittent intravenous bolus or intravenous continuous infusion of cefotaxime in critically ill patients. Critically ill patients will be randomized to intermittent infusion or continuous infusion of cefotaxime.

DETAILED DESCRIPTION:
Critically ill patients have other pharmacokinetic/pharmacodynamic profiles than healthy volunteers. Suboptimal, both under- and overdosing of antibiotics is an important threat in this patient category. Given the time-dependent character of beta-lactam antibiotics continuous dosing as opposed to traditional intermittent dosing is likely to render better target attainment and maintenance and might improve clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care
* Able to give informed consent by themselves or informed consent can be obtained via next of kin
* Indication for treatment with cefotaxime (as judged by treating physician) in the context of our standard treatment protocol of Selective decontamination of the digestive tract (SDD).

Exclusion Criteria:

* Renal replacement therapy
* Contra-indication for cefotaxime, including known or suspected allergy to cefotaxime
* No indication for an arterial line; an arterial line will not be placed solely for the purpose of this study; thus, only patients with an indication for an arterial line outside this protocol are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cefotaxim serum concentrations | 40 min, 1 hour, 2, 4, 8, 12 and 24 hours; 36h; 48 h; 60h; 72h; 84h and 96h post administration
  Cefotaxime serum concentrations, total and unbound, will be determined. The Pharmacokinetic/Pharmacodynamic (PK/PD) target of total serum concentration of 4 times above minimal inhibitory concentration (MIC) ascertains that the unbound drug serum concentration will be above the MIC value of 1 mg/mL, which is determined to be the minimum target.

SECONDARY OUTCOMES:
Area under the curve of cefotaxim | 0-96h post administration
  Based on the data from the primary outcome measure a pharmacokinetic model for ICU patients will be developed.

CONTACTS AND LOCATIONS:
Overall Officials: Jan G Zijlstra, MD, PhD, Principal Investigator — Department of Critical Care, UMCG
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Aardema H, Bult W, van Hateren K, Dieperink W, Touw DJ, Alffenaar JC, Zijlstra JG. Continuous versus intermittent infusion of cefotaxime in critically ill patients: a randomized controlled trial comparing plasma concentrations. J Antimicrob Chemother. 2020 Feb 1;75(2):441-448. doi: 10.1093/jac/dkz463. PMID 31697336